CLINICAL TRIAL: NCT05372965
Title: The Effects of Smoking on miRNA-223 Before and After Non-Surgical Periodontal Therapy
Brief Title: The Effects of Smoking on miRNA-223 Before-After Non-Surgical Periodontal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Burcu KARADUMAN, Doç. Dr., Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2015-KAEK-58-22-02
Record Dates: First submitted 2022-04-29; First posted 2022-05-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Periodontal Therapy; miRNA-223; Periodontitis; Biomarker
Keywords: periodontal therapy; biomarker; periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Our study will include 42 people with periodontitis and 42 healthy periodontal patients (84 individuals in total), and these two groups will be divided into two as smokers and non-smokers. Clinical measurements (Plaque index, probing depth, gingival recession, clinical attachment level, bleeding on probing) and salivary sample will be taken from all individuals at the beginning of the study. Non-surgical periodontal treatment will be applied to individuals with periodontitis, gingival samples will be collected during the treatment, clinical measurements and saliva collection will be repeated 6 weeks after the treatment. MiRNA-223 gene expression analysis will be performed by real-time PCR method in saliva and gingival samples of individuals. MiRNA-223 and cotinine levels will be examined to evaluate the effects of smoking before and after treatment in periodontal health and periodontitis.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: periodontitis (Experimental): Our study will include 42 people with periodontitis patients and these two groups will be divided into two as smokers (21) and non-smokers (21).
  Interventions: Other: experimental-periodontitis-mirna-223-gingival tissue-saliva samples
- Control: clinical healthy (Active Comparator): Our study will include 42 people with clinical healthy patients and these two groups will be divided into two as smokers (21) and non-smokers (21).
  Interventions: Other: control-clinical healthy mirna-223-gingival tissue-saliva samples

INTERVENTIONS:
Other: experimental-periodontitis-mirna-223-gingival tissue-saliva samples — Non-surgical periodontal treatment will be applied to individuals with periodontitis, gingival samples will be collected during the treatment, clinical measurements and saliva collection will be repeated 6 weeks after the treatment. MiRNA-223 gene expression analysis will be performed by real-time PCR (Polymerase Chain Reaction) method in saliva and gingival samples of individuals. MiRNA-223 and cotinine levels will be examined to evaluate the effects of smoking before and after treatment in periodontal health and periodontitis. Clinical measurements (Plaque index, probing depth, gingival recession, clinical attachment level, bleeding on probing) and salivary sample will be taken from all individuals at the beginning of the study.
  Arms: Experimental: periodontitis
Other: control-clinical healthy mirna-223-gingival tissue-saliva samples — Clinical measurements (Plaque index, probing depth, gingival recession, clinical attachment level, bleeding on probing) and salivary sample will be taken from all individuals at the beginning of the study. MiRNA-223 and cotinine levels will be examined to evaluate the effects of smoking before and after treatment in periodontal health and periodontitis. A pre-treatment saliva sample will be collected from the clinically healthy group. A tissue sample will be collected during the clinical crown lengthening operation.
  Arms: Control: clinical healthy

SUMMARY:
Periodontal diseases are one of the most common inflammatory diseases. Periodontal disease results from a complex interplay between the subgingival biofilm and the host immune-inflammatory events that develop in the gingival and periodontal tissues in response to the challenge presented by the bacteria. The net result of these inflammatory changes is the breakdown of the fibers of the periodontal ligament, resulting in clinical loss of attachment together with resorption of the alveolar bone. It is known that smoking is a major risk factor for periodontitis and affects the occurrence and severity of the disease and recovery after periodontal treatment by changing the host response to plaque. Biomarkers can be used to diagnose periodontitis early, to determine the rate of destruction, and also to evaluate the response to treatment. It has been reported that microRNAs (miRNAs) play an important role in development, homeostasis and immune functions, and abnormal miRNA expression may increase the severity of disease progression. It can be thought that early diagnosis can be achieved with the detection of miRNAs in patients with periodontitis, thus helping to prevent bone and tooth loss. To the best of our knowledge, there is no study in the literature investigating the effects of periodontal treatment and smoking on miRNAs in saliva or gingival samples. From this point of view, the aim of our study is to examine and compare miRNA-223 expressions in saliva and tissue samples before and after non-surgical periodontal treatment in individuals with periodontitis and to investigate the effect of smoking on miRNA-223 levels.

Materials-Methods: Our study will include 42 people with periodontitis and 42 healthy periodontal patients (84 individuals in total), and these two groups will be divided into two as smokers and non-smokers. Clinical measurements (Plaque index, probing depth, gingival recession, clinical attachment level, bleeding on probing) and salivary sample will be taken from all individuals at the beginning of the study. Non-surgical periodontal treatment will be applied to individuals with periodontitis, gingival samples will be collected during the treatment, clinical measurements and saliva collection will be repeated 6 weeks after the treatment. MiRNA-223 gene expression analysis will be performed by real-time PCR method in saliva and gingival samples of individuals. MiRNA-223 and cotinine levels will be examined to evaluate the effects of smoking before and after treatment in periodontal health and periodontitis.

With our study, it is aimed to better illuminate the role of miRNA-223 in periodontitis and also to determine which sample is more reliable by comparing miRNA-223 levels in saliva and tissue samples. Thus, the first step towards the development of diagnostic kits in the future will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Periodontal healthy group
* Stage III Grade B-C Periodontitis Group
* To meet the above-mentioned periodontal health and disease criteria

Exclusion Criteria:

* Periodontal tissues, periodontal disease course, periodontal application training and to have,
* Chronic alcohol use,
* Oral contraceptive use, pregnancy, pregnant,
* Last 6 system or anti-inflammatory drug use,
* To have developed periodontal in the last 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Examination of miRNA-223 expressions, which are stated to be associated with periodontal disease, in saliva and gingival samples obtained from individuals with periodontitis, | During study (up to 1 year)
  With our study, it is aimed to better illuminate the role of miRNA-223 in periodontitis and also to determine which sample is more reliable by comparing miRNA-223 levels in saliva and tissue samples. Thus, the first step towards the development of diagnostic kits in the future will be taken.
Evaluation of the effect of non-surgical periodontal treatment on changes in miRNA-223 expressions, | 6 weeks after the non surgical periodontal therapy
  Non-surgical periodontal treatment will be applied to individuals with periodontitis, gingival samples will be collected during the treatment, clinical measurements and saliva collection will be repeated 6 weeks after the treatment.
Examining the effect of smoking, which is one of the main risk factors of periodontitis, on miRNA-223 levels and | through study completion, an average of 1 year
  the aim of our study is to examine and compare miRNA-223 expressions in saliva and tissue samples before and after non-surgical periodontal treatment in individuals with periodontitis and to investigate the effect of smoking on miRNA-223 levels.

SECONDARY OUTCOMES:
to determine which sample is more reliable by comparing miRNA-223 levels in saliva and tissue samples | through study completion, an average of 1 year
  With our study, it is aimed to better illuminate the role of miRNA-223 in periodontitis and also to determine which sample is more reliable by comparing miRNA-223 levels in saliva and tissue samples. Thus, the first step towards the development of diagnostic kits in the future will be taken.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni Üniversitesi, Istanbul, İstanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided